CLINICAL TRIAL: NCT00915200
Title: N-Acetylcysteine and Milk Thistle for Treatment of Diabetic Nephropathy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NIH 1R21AT004490; 1I01CX000264-01A2 (NIH); R21AT004490 (NIH)
Record Dates: First submitted 2009-06-02; First posted 2009-06-05 (Estimated); Last update posted 2016-06-27 (Estimated); Status verified 2016-06

CONDITIONS: Diabetic Nephropathies; Proteinuria; Oxidative Stress
Keywords: Diabetic Nephropathies; Proteinuria; Renal Insufficiency, Chronic; Monocytes; Oxidative stress; Inflammation; Antioxidants; Glutathione; Silymarin; Acetylcysteine; Dietary Supplements; Complementary Therapies
MeSH Terms: conditions — Diabetic Nephropathies; Proteinuria; Renal Insufficiency, Chronic; Inflammation | interventions — Acetylcysteine; Silybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): N-acetylcysteine placebo + silibin placebo
  Interventions: Dietary Supplement: N-acetylcysteine placebo; Dietary Supplement: silibin placebo
- N-acetylcysteine (Experimental): N-acetylcysteine active + silibin placebo
  Interventions: Dietary Supplement: N-acetylcysteine; Dietary Supplement: silibin placebo
- silibin (Experimental): N-acetylcysteine placebo + silibin active
  Interventions: Dietary Supplement: silibin; Dietary Supplement: N-acetylcysteine placebo; Dietary Supplement: silibin placebo
- N-acetycysteine + silibin (Experimental): N-acetylcysteine active + silibin active
  Interventions: Dietary Supplement: N-acetylcysteine; Dietary Supplement: silibin; Dietary Supplement: silibin placebo
- N-acetylcysteine + high-dose silibin (Experimental): N-acetylcysteine active + high-dose silibin active
  Interventions: Dietary Supplement: N-acetylcysteine; Dietary Supplement: high-dose silibin

INTERVENTIONS:
Dietary Supplement: N-acetylcysteine — 600 mg orally twice daily for three months
  Other Names: NAC
  Arms: N-acetycysteine + silibin; N-acetylcysteine; N-acetylcysteine + high-dose silibin
Dietary Supplement: silibin — 480 mg orally twice daily for three months
  Other Names: silibin-phosphatidylcholine, Siliphos
  Arms: N-acetycysteine + silibin; silibin
Dietary Supplement: high-dose silibin — 960 mg orally twice daily for three months
  Other Names: silibin-phosphatidylcholine, Siliphos
  Arms: N-acetylcysteine + high-dose silibin
Dietary Supplement: N-acetylcysteine placebo — excipient orally twice daily for three months
  Other Names: NAC placebo
  Arms: Placebo; silibin
Dietary Supplement: silibin placebo — excipient orally twice daily for three months
  Other Names: silibin-phosphatidylcholine placebo, Siliphos placebo
  Arms: N-acetycysteine + silibin; N-acetylcysteine; Placebo; silibin

SUMMARY:
The study is designed to test if the combination of two potent antioxidant nutritional supplements, N-acetylcysteine and the milk thistle extract silibin, is capable of correcting the shedding of urine protein, the oxidative stress, and the inflammation in patients with type 2 diabetes mellitus and diabetic kidney disease.

DETAILED DESCRIPTION:
Oxidative stress and GSH imbalance are major contributors to the pathogenesis of diabetic nephropathy. Current options for the treatment of oxidative stress in diabetic nephropathy are limited and only partially effective, thus interest in the development of new strategies is high.

The study intends to test the hypothesis that combined oral supplementation of the antioxidants N-acetylcysteine (NAC) and milk thistle flavonolignan silibin (as silibin-phosphatidylcholine) will reduce proteinuria and urinary and systemic manifestations of oxidative stress and inflammation, which are characteristically observed in patients with type 2 diabetes mellitus and related nephropathy. We expect these effects to be achieved with minimal or no side effects, and with good patient tolerance.

The trial is designed as a two-center, double-blind, placebo-controlled, randomized, modified-factorial dose-ranging design, five-arm pilot study in patients with Type 2 diabetes mellitus and advanced diabetic nephropathy with proteinuria.

Intervention consists of three-month oral administration of NAC, silibin, and/or respective placebos for three months. Subjects are randomized to the following five intervention arms: (A) placebo; (B) NAC; (C) silibin; (D) NAC + silibin; and (E) NAC + double-dose silibin.

The primary outcome measure is urinary excretion of albumin, a marker of glomerular injury. Secondary outcome measures are alpha-1 microglobulin, a marker of tubular injury, and urinary excretion of inflammatory cytokines and C-C chemokines, i.e. markers of renal inflammation. In addition, peripheral blood monocytes from the same patients are analyzed for glutathione (GSH) content and activity of GSH metabolizing enzymes. All outcome measures are monitored in relation to both treatment allocation and prevalent blood and urine levels of the active treatment. Safety and tolerability of this combination treatment are monitored throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Males or females, age 18-70 years old.
* Type 2 diabetes mellitus
* Diabetic nephropathy, as defined by:

  * estimated GFR between 60 and 15 ml/min,
  * presence of proteinuria.
* Current medical treatment with low dose aspirin
* Treatment of hypertension with (but not limited to) one diuretic, one beta- blocker and one medication from the classes ARBs or ACE inhibitors.
* Treatment of hyperglycemia with (but not limited to) glipizide and the medication class insulin.
* Treatment of hypercholesterolemia with (but not limited to) one medication from the class statins.

Exclusion Criteria:

* Type 1 diabetes mellitus.
* Glycosylated hemoglobin (HbA1C) > 10%
* >20% variation in estimated GFR, during last 6 months
* SBP >170 mmHg or DBP >100 mmHg on medications
* Other secondary forms of hypertension (endocrine, renovascular)
* History of intolerance to:

  * Both ACE-I and ARBs;
  * The investigational supplements;
  * Iodinated radiologic contrast material.
* Known non diabetic renal disease, or history of solid organ transplantation.
* Hepatitis virus or Human Immunodeficiency virus infections
* Use of one of the following medications within 2 months prior to enrollment in the study:

  * Metformin.
  * Thiazolidinediones (pioglitazone or rosiglitazone);
  * Prescription-grade vitamin E, vitamin C, systemic steroids, and/or non-steroidal anti-inflammatory agents;
  * Over-the-counter vitamin E, vitamin C, and/or non-steroidal anti-inflammatory agents.
  * Over-the-counter antioxidants supplements including: Lipoic acid, Coenzyme Q10, N-acetyl-cysteine (NAC), Glutathione (GSH), Chromium, Fish-oil extracts (omega-3 fatty acids), Soy extracts (isoflavones), Milk thistle extract (silymarin), Green-tea preparations, Pomegranate extracts, Grape extracts, and Prickly pear extract.
* Active coronary artery disease or cerebral vascular disease within 3 months prior to signing the informed consent.
* Hepatic dysfunction as defined by abnormal total bilirubin or liver enzymes (ALT, AST) >2 times upper limit of normal range.
* Active malignancy.
* History of drug or alcohol dependency.
* Psychiatric or neurological condition, preventing aware consent to the study and/or adherence to the study protocol
* Unwillingness to practice birth control throughout the study.
* Participation to another clinical study within 1 month prior to signing the informed consent form.
* Planned move to outside the study area, surgery or radiographic studies utilizing iodine-based contrast material within the next one year

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2009-10; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Urinary Albumin excretion | 3-month

SECONDARY OUTCOMES:
urinary alpha-1 microglobulin excretion | 3-month
urinary C-C-chemokines excretion | 3-month
peripheral blood monocyte glutathione content | 3-month
tolerance and safety | 3-month

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Fanti, M.D., Principal Investigator — University of Texas
Locations (1):
- University of Texas Hlth Sci Ctr San Ant, San Antonio, Texas, United States

REFERENCES:
- [Derived] Colombijn JM, Hooft L, Jun M, Webster AC, Bots ML, Verhaar MC, Vernooij RW. Antioxidants for adults with chronic kidney disease. Cochrane Database Syst Rev. 2023 Nov 2;11(11):CD008176. doi: 10.1002/14651858.CD008176.pub3. PMID 37916745